CLINICAL TRIAL: NCT03678714
Title: Effects of Exercise on Oxidised LDL and Cardiometabolic Profile in Women With Polycystic Ovary Syndrome: Study Protocol for a Feasibility Randomized-controlled Trial
Brief Title: Effect of Exercise on Cardiometabolic Profile in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ER6262197
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; exercise; physical activity; cardiovascular disease; low-density lipoprotein; metabolism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomised into either an exercise group, a lifestyle physical activity group, or a control group, for a duration of 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to mask participants or research team to the allocated intervention. Outcome assessors will be blinded to group allocation for anthropometric and fitness measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Intervention (Experimental): Structured exercise intervention will be undertaken for 12 weeks
  Interventions: Behavioral: Exercise Intervention
- Lifestyle Physical Activity (Experimental): Increased lifestyle physical activity undertaken for 12 weeks
  Interventions: Behavioral: Lifestyle Physical Activity
- Control (No Intervention): Resting control

INTERVENTIONS:
Behavioral: Exercise Intervention — 2 sessions of supervised exercise training each week for 8 consecutive weeks and 3 sessions of supervised exercise training each week for the final 4 consecutive weeks, at 57-74% heart-rate max. Each session will last approximately 60 minutes.
  Arms: Exercise Intervention
Behavioral: Lifestyle Physical Activity — Advice and information on how to increase physical activity will be provided. Participants will be asked to monitor and track their daily physical activity using a smart-phone fitness application. The research team will gain permission to access their recorded activity.
  Arms: Lifestyle Physical Activity

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is a complex hormonal and metabolic disorder that has been shown to affect women's fertility. It can also share many symptoms with pre-diabetes, and women with PCOS often have an increased risk for type 2 diabetes, heart attack and stroke.

This study aims to assess the feasibility and acceptability of exercise intervention and increased lifestyle physical activity to improve cardiovascular disease risk factors in women with PCOS.

DETAILED DESCRIPTION:
This is a three arm feasibility study in which participants will be allocated to an exercise group, an increased lifestyle physical activity group, or a control group. We will determine the appropriateness of procedures for recruitment, allocation, measurement and retention for the intervention procedures in women with polycystic ovary syndrome.

The investigators will also determine if we are able to detect changes in blood lipid profile, inflammation, and hormonal and metabolic profile as a result of the intervention(s) using blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS according to the Rotterdam Criteria 2003, National Institute of Health (NIH) 1990 criteria or Androgen Excess and Polycystic Ovary Syndrome (AE-PCOS) Society 2006 criteria.
* Have experienced menarche (their first menstrual bleeding) and be at least 18 years of age.
* Are English speaking.
* Are physically able to perform exercise.

Exclusion Criteria:

* Post-menopausal status.
* Are smokers.
* Are undertaking regular structured exercise defined as >150min/week.
* Have been taking metformin for less than three months.
* Are taking the oral contraceptive pill (OCP) or have taken in the last month.
* Have any medical condition that may be responsible for the symptoms of PCOS, such as congenital hyperplasia, androgen-secreting tumour, hyperprolactinemia, or Cushing's syndrome.
* Have current cardiovascular disease or a history of cardiac events.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | One year
  Recruitment rate will be calculated by dividing the number of women eligible and consenting by the recruitment period.
Attrition Rate | One year
  Attrition rates will be established as discontinuation of the intervention and loss to follow-up measurement for both conditions.
Compliance to intervention | One year
  Compliance will be monitored by session attendance and monitoring the data from recorded daily physical activity, with examination of reasons for drop-out or non-compliance
Suitability of allocation and measurement procedures | One year
  Reasons for drop-out will be used to assess the suitability of allocation procedures. Suitability of measurement procedures will be evaluated by completion rates and reasons for missing data.

SECONDARY OUTCOMES:
Oxidised low-density lipoprotein mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
Free testosterone mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
Fasting insulin mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
C-reactive protein mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
Thiobarbituric Acid and Reactive Substances (TBARS) mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
Neopterin mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
Sex hormone binding globulin mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
High density lipoprotein cholesterol mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
Low density lipoprotein cholesterol mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
Triglycerides mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
Total cholesterol mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks
Fasting glucose mean change from baseline | Baseline and 12-weeks
  Blood samples are taken from all participants at baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amie Woodward, MSc, Principal Investigator — Sheffield Hallam University; Markos Klonizakis, PhD, Study Director — Sheffield Hallam University
Locations (1):
- Centre for Sports and Exercise Science, Sheffield Hallam University, Sheffield, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Woodward A, Broom D, Dalton C, Metwally M, Klonizakis M. Supervised exercise training and increased physical activity to reduce cardiovascular disease risk in women with polycystic ovary syndrome: study protocol for a randomized controlled feasibility trial. Trials. 2020 Jan 20;21(1):101. doi: 10.1186/s13063-019-3962-7. PMID 31959233